CLINICAL TRIAL: NCT01268137
Title: DEEP BRAIN STIMULATION IN TREATMENT RESISTANT MAJOR DEPRESSION. Controlled and Crossed Study on Efficacy and Safety.
Brief Title: DBS in Treatment Resistant Major Depression
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Collaborators: Fondo de Investigacion Sanitaria (Other)
Responsible Party: Jordi Virgili, Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: DEP-012004
Record Dates: First submitted 2010-12-28; First posted 2010-12-29 (Estimated); Last update posted 2010-12-29 (Estimated); Status verified 2010-12

CONDITIONS: Resistant Major Depressive Disorder
Keywords: MDD; DBS
MeSH Terms: interventions — Deep Brain Stimulation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- stimulation on (Active Comparator): At first stage, electrodes will be implanted in all patients, who will be continuously stimulated for several months. After this stage, the random-crossed part of the study will start, and patients who responded to DBS will be randomly distributed in two groups: on stimulation or off stimulation group, for the next three months. Subsequently, patients will be allocated in the other group (on or off, crossed part) for three months
  Interventions: Procedure: Deep Brain Stimulation
- Stimulation off (Placebo Comparator): At first stage, electrodes will be implanted in all patients, who will be continuously stimulated for several months. After this stage, the random-crossed part of the study will start, and patients who responded to DBS will be randomly distributed in two groups: on stimulation or off stimulation group, for the next three months. Subsequently, patients will be allocated in the other group (on or off, crossed part) for three months
  Interventions: Procedure: Deep Brain Stimulation

INTERVENTIONS:
Procedure: Deep Brain Stimulation — Surgical electrode implantation in the white matter adjacent to the Cg25 region and implantation of the DBS pulse generating device

SUMMARY:
This study aims at assessing efficacy and safety of DBS for treatment of patients suffering from resistant major depression, by means of a random, controlled and crossed study.

DETAILED DESCRIPTION:
The first phase of the study will consist of implanting electrodes and applying continuous stimulation until the patients stabilise clinically. This period is anticipated between 6 and 9 months. The next phase will consist of the crossover study. Responders will be randomised to either of 2 groups for a period of 3 months: a stimulation-on group and a stimulation-off group. Patients will then be crossed over to the other group for a further 3 months. Fortnightly visits will be made during the entire study to evaluate treatment efficacy and patient tolerance

ELIGIBILITY:
Inclusion Criteria:

1. Patients of both sexes aged between 18 and 70 years.
2. Patients diagnosed as having an MDD episode according to DSM-IV-TR criteria, resistant to pharmacological treatment with a score of 4 in the Thase-Rush index, with ECT contraindicated or having failed to produce a maintained response.
3. Patients with a HRSD-17 score of 18 or more.
4. Patients with an intellectual capacity that facilitates adequate communication and who are willing to cooperate with all the examinations and protocols of the study.
5. Patients who have not modified their antidepressant treatment in the month prior to the study.
6. Women of childbearing age using medically approved contraceptive methods.
7. Patients who have granted their informed consent in writing.

Exclusion Criteria:

1. Female patients who are pregnant or breastfeeding.
2. Patients with acute, serious or unstable illnesses.
3. Patients experiencing delirium or hallucinations, congruent or otherwise with their mood.
4. Patients with a history of substance abuse (other than tobacco or caffeine).
5. Patients with concomitant psychiatric disorders from axes I or II of DSM IV-TR.

h)Patients with general contraindications for DBS (pacemaker users, etc).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2008-01; Primary Completion 2011-06 (Estimated); Study Completion 2011-06 (Estimated)

PRIMARY OUTCOMES:
Hamilton Rating Scale for Depression, 17-item version (HRSD-17) | Psychiatric assessments will be performed every two weeks

SECONDARY OUTCOMES:
Montgomery-Asberg Depression Rating scale (MADRS) Clinical Global Impression (CGI) of Severity/Improvement Neuropsychological variables | Psychiatric assessments will be performed every two weeks

CONTACTS AND LOCATIONS:
Overall Officials: Perez Sola Víctor, MD, Principal Investigator — Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau; Molet Joan, MD, Principal Investigator — Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau
Locations (1):
- Hospital Santa Creu i Sant Pau, Barcelona, Spain

REFERENCES:
- [Derived] Puigdemont D, Portella M, Perez-Egea R, Molet J, Gironell A, de Diego-Adelino J, Martin A, Rodriguez R, Alvarez E, Artigas F, Perez V. A randomized double-blind crossover trial of deep brain stimulation of the subcallosal cingulate gyrus in patients with treatment-resistant depression: a pilot study of relapse prevention. J Psychiatry Neurosci. 2015 Jul;40(4):224-31. doi: 10.1503/jpn.130295. PMID 25652752
- [Derived] Puigdemont D, Perez-Egea R, Portella MJ, Molet J, de Diego-Adelino J, Gironell A, Radua J, Gomez-Anson B, Rodriguez R, Serra M, de Quintana C, Artigas F, Alvarez E, Perez V. Deep brain stimulation of the subcallosal cingulate gyrus: further evidence in treatment-resistant major depression. Int J Neuropsychopharmacol. 2012 Feb;15(1):121-33. doi: 10.1017/S1461145711001088. Epub 2011 Jul 22. PMID 21777510